CLINICAL TRIAL: NCT01944228
Title: Effects of Transvenous Vagus Nerve Stimulation on Immune Response: a Pilot Study
Acronym: NoSIRS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NoSIRS Study; 2012-005687-97 (EudraCT Number)
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Inflammation
Keywords: inflammation; vagus nerve stimulation; chronic heart failure; Systemic Inflammatory Response Syndrome; sepsis; auto-immune diseases
MeSH Terms: conditions — Inflammation; Systemic Inflammatory Response Syndrome; Sepsis | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vagal Nerve Stimulation (Experimental): 30 minutes of vagal nerve stimulation using a catheter in the IJV
  Interventions: Device: Vagal Nerve Stimulation
- Sham stimulation (Sham Comparator): Catheter placed in the IJV without stimulation
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: Vagal Nerve Stimulation — 30 minutes of vagal nerve stimulation using a catheter in the IJV
  Arms: Vagal Nerve Stimulation
Device: Sham Stimulation — Catheter placed in the IJV without stimulation
  Arms: Sham stimulation

SUMMARY:
The purpose of this study is to assess the effect of transvenous vagus nerve stimulation (tVNS) on the immune response.

In the human endotoxemia model, intravenously administered endotoxin (lipopolysaccharide [LPS]) elicits a systemic immune response with release of pro-inflammatory cytokines, such as TNF α. This trial will determine if an anti-inflammatory effect can be produced by acute VNS using a minimally invasive delivery method.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent to participate in this trial
2. Male subjects aged 18 to 35 years inclusive
3. Healthy as determined by medical history, physical examination, vital signs, 12 lead electrocardiogram, and clinical laboratory parameters

Exclusion Criteria:

* Use of any medication(including herbal remedies and vitamin/mineral supplements) or recreational drugs within 7 days prior to profiling day
* Smoking
* Use of caffeine, or alcohol or within 1 day prior to profiling day
* Previous participation in a trial where LPS was administered
* Surgery or trauma with significant blood loss or blood donation within 3 months prior to profiling day
* Participation in another clinical trial within 3 months prior to profiling day.
* History, signs or symptoms of cardiovascular disease
* An implant that in the opinion of the investigator may make invasive procedures risky for the subject due to the increased risks associated with a possible infection.
* Subject has an implanted active cardiac device (ICD, IPG and/or CRT)
* Implanted active neurostimulation device
* Subject has internal jugular vein that cannot be accessed
* History of vaso-vagal collapse or of orthostatic hypotension
* History of atrial or ventricular arrhythmia
* Resting pulse rate ≤45 or ≥100 beats / min
* Hypertension (RR systolic >160 or RR diastolic >90)
* Hypotension (RR systolic <100 or RR diastolic <50)
* Conduction abnormalities on the ECG consisting of a 1st degree atrioventricular block or a complex bundle branch block
* Subject is diagnosed with epilepsy or history of seizures
* Renal impairment: plasma creatinine >120 µmol/L
* Liver function abnormality: alkaline phosphatase>230 U/L and/or ALT>90 U/L
* Coagulation abnormalities: APTT or PT > 1.5 times the reference range
* History of asthma
* Immuno-deficiency
* CRP > 20 mg/L, WBC > 12x109/L, or clinically significant acute illness, including infections, within 2 weeks before profiling day
* Known or suspected of not being able to comply with the trial protocol
* Inability to personally provide written informed consent (e.g. for linguistic or mental reasons) and/or take part in the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2013-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Plasma TNF-α concentration | 24 hours
  Plasma TNF-α concentration after LPS administration (Area Under Curve); comparison of subjects treated with tVNS versus sham tVNS.

SECONDARY OUTCOMES:
Plasma concentrations of pro-inflammatory and anti-inflammatory cytokines | up to 24 h
  Plasma concentrations of pro-inflammatory and anti-inflammatory cytokines (including TNF-α, IL 6, IL 1RA, IL 10) up to 24 h after LPS injection to document the immune response up to 24 hrs; comparison of subjects treated with tVNS versus sham tVNS.
Leukocyte responses to ex vivo stimulation | up to 24 hrs
  Leukocyte responses to ex vivo stimulation with inflammatory stimuli and leukocyte phagocytosis capacity up to 24 hrs; comparison of subjects treated with tVNS versus sham tVNS
Endotoxemia-related clinical symptoms | up to 24 hrs
  Endotoxemia-related clinical symptoms, hemodynamic parameters, and temperature up to 24 hrs; comparison of subjects treated with tVNS versus sham tVNS.
Endotoxemia-induced circulating leukocyte changes | up to 24 hrs
  Endotoxemia-induced circulating leukocyte changes up to 24 hrs; comparison of subjects treated with tVNS versus sham tVNS.
Autonomic nervous system activity | up to 24 hrs
  Autonomic nervous system activity measured by heart rate variability up to 24 hrs; comparison of subjects treated with tVNS versus sham tVNS.
Tolerability of acute side effects of tVNS | Acute 30 min stimulation
  Tolerability of acute side effects of tVNS. Subject feedback during VNS.
Ease of tVNS delivery | acute interoperative
  Perception of delivery difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pickkers, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] Kox M, van Eijk LT, Verhaak T, Frenzel T, Kiers HD, Gerretsen J, van der Hoeven JG, Kornet L, Scheiner A, Pickkers P. Transvenous vagus nerve stimulation does not modulate the innate immune response during experimental human endotoxemia: a randomized controlled study. Arthritis Res Ther. 2015 Jun 7;17(1):150. doi: 10.1186/s13075-015-0667-5. PMID 26049730